CLINICAL TRIAL: NCT03334045
Title: Neurobiological Effects of Work-related Adjustment Disorder
Acronym: NeuroWAD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Saga Steinmann Madsen, Clinical Engineer, Odense University Hospital
Other Study IDs: OP_483
Record Dates: First submitted 2017-10-13; First posted 2017-11-07 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Adjustment Disorder With Work Inhibition
Keywords: Neurobiology; Occupational Stress; Dopamine
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stress patients: Patients diagnosed with work-related Adjustment disorder
  Interventions: Radiation: PET/MR scans
- Controls: Healthy controls
  Interventions: Radiation: PET/MR scans

INTERVENTIONS:
Radiation: PET/MR scans — Observations of glucose metabolism and dopamine binding potential

SUMMARY:
INTRODUCTION: Stress is one of the greatest burdens of our society and often imply impairments in cognitive and emotional functions. The investigators hypothesize that changes in the brain's dopamine(DA)-based mesocorticolimbic projections in patients with work-related stress (adjustment disorder) will manifest in altered glucose metabolism in relation to neural activity and altered DA radiotracer binding potential at neurotransmitter and receptor level.

MATERIAL AND METHODS: Subjects and healthy controls undergo neuropsychiatric tests and PET/MR imaging with three tracers: [18F]FDG to measure glucose metabolism as a marker of neural activity, [11C]raclopride to investigate the DA binding potential in the striatum, and [11C]FLB 457 to study possible impaired mesocortical dopaminergic transmission. To demonstrate difference in glucose metabolism ≥2x41 patients/controls are needed.

OUTCOME: The investigators expect to find that symptoms of cognitive and motivational/reward deficits could be attributable to changes in frontal lobe and striatal glucose metabolism in >50% of patients and that changes in striatal D2 receptors and impaired mesocortical dopaminergic transmission in the prefrontal cortex are contributing factors.

CONCLUSION: This project aims to generate entirely new and objective evidence of stress-induced cerebral illness and provide a basis for in depth research and more rational management of this strenuous disorder.

DETAILED DESCRIPTION:
Recruitment procedure: The department of Occupational and Environmental Medicine (DOE) at OUH have developed a screening procedure to recruit patients diagnosed according to the ICD10 F43.2x, and exposed to predominant psychosocial work stressors. The patients are recruited among women and men aged 18-64. At the DOE subjects undergo a clinical diagnostic interview based on the ICD 10 criteria including screening for stressors in the psychosocial work environment and their relationship to disease development, private life strains, personal back-ground, mental vulnerability, and competing somatic disease, as well as tests for depression and anxiety symptoms, respectively the Beck Anxiety Inventory (BAI) and Major Depression Inventory (MDI). The psychosocial work environ-ment stressors being screened for are: quantitative demands, emotional demands, role conflict, role ambiguity, sup-port and encouragement, organizational justice, adequate education and training (skill level). The experience of stressors is assessed in relation to the most dominant stress models, "demand-control-support" (Karasek), "effort and reward imbalance at work" (Siegrist), "Stress as Offense two self" (Semmer), and classical stress theory focusing on appraisal / coping (Lazarus or Ursin).

The procedure is onward going to be performed automatically in an online environment. Due to the nature of neurobiology the scans must be conducted within a fairly short time period after the initial diagnosis. Hence a declaration of consent will be presented and signed at the day of the first scan, also ensuring that all additional questions can be answered by the main investigator. The scans will be conducted within a fortnight after the fists contact. In connection with the scans, the main investigator will conduct an SCAN-PSE interview for the assessment of mental symptoms to determine if the participant's condition has changed since they decided to participate in the trial. Healthy controls are recruited and matched with regard to gender, age, educational and occupational background. Further, controls are screened for confounding factors in a similar manner as the patient group.

ELIGIBILITY:
Inclusion Criteria:

Population and controls:

* Informed consent before study-related activity
* Aged 18 - 64
* Labour market suitability

Study population:

* Patients: F43.2
* Controls: Healthy individuals that meet the following inclusion and

Exclusion criteria.

Population, patients and controls:

* Comorbid diagnoses as for instance: cancer, cardiovascular disease, diabetes.
* Regular medication known to affect the central nervous system.
* Prior exposure to violence and other serious harassment in the workplace
* Psychosocial challenge in private life according to the screening criteria in the protocol.
* Other serious illness
* Metal in body
* Claustrophobia
* Pregnancy
* Confounding drug consumption
* Dependence e.g. alcohol, narcotics or other
* Persons within a period of 1 year have participated in scientific studies that use isotopes, or who have had greater diagnostic tests that utilize ionizing radiation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The patients are recruited among women aged 18-64 years.
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Glucose metabolism | 3 year
  PET/MR scan

SECONDARY OUTCOMES:
Dopamine binding potential | 3-4 years
  PET/MR scan

CONTACTS AND LOCATIONS:
Overall Officials: Saga Steinmann Madsen, Engineering, Principal Investigator — OUH
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madsen SS, Gjedde A, Brandt L, Pihl-Thingvad J, Videbech P, Gerke O, Hojlund-Carlsen PF. Neurobiological effects of work-related stress: protocol for a case-control neuroimaging study. Dan Med J. 2018 Nov;65(11):A5513. PMID 30382017